CLINICAL TRIAL: NCT05811338
Title: Center for Research and Education on Aging and Technology Enhancement - CREATE V
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-01025559; P01AG073090-01A1 (NIH)
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Technology
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Project 1 - Phase 1: Development/Refinement of VR program; Usability Testing/Development of Training (No Intervention): The study includes one session that will last approximately 2 - 3 hours. The study involves completing some questionnaires that gather background demographic information and a structured needs assessment interview to gather information on user preferences, usability problems, implementation and training protocols.
- Project 1 - Phase 2: VR Program (Experimental): Training will occur over 3 days and be conducted by research investigators in the participants' homes. Training will include training on the proper placement of the headset, the viewing lens, system headphones, and safety guidelines. The research investigator will aid in the set-up of the VR system in the home, which will be pre-loaded with applications, and will recommend an area to use the system to ensure a safe play area free of obstacles. Participants will be provided with practice tasks between training sessions. Participants will be provided with a "hands-on" performance assessment at the beginning of the second session and concepts/procedures that are problematic will be reviewed. Participants will be contacted one-week post training to determine if they are having any problems by study investigators. Following training, participants will use the CAST VR program and tablet at will, though encouraged to use it at least three times per week for 20 minutes.
  Interventions: Behavioral: Project 1, Phase 2: VR Program for Social, Activity, and Cognitive Engagement
- Project 1 - Phase 2: Tablet Control Condition (Active Comparator): Training will occur over 3 days and be conducted by research investigators in the participants' homes. Participants in the control condition will receive a tablet, internet support for 2 months and training (including training on cybersecurity). This will include instructions for accessing content similar to, but in 2-D, so less immersive than that included in the VR program (e.g., virtual museum tours, One click, etc.). Participants will complete all assessments and will be provided with an Android tablet that has a 10.1" display, built in modem, and a front facing camera. Research investigators are providing people with tablets for standardization. Research Assessor (RA) Training, Certification and Treatment Fidelity. At follow-up assessments, assessors and data analysts will be blinded to treatment condition.
  Interventions: Behavioral: Project 1, Phase 2: VR Program for Social, Activity, and Cognitive Engagement
- Project 2 - Phase 2: Active Intervention Group (Experimental): Participants will receive a tablet with the adaptive program and be provided with internet service following the baseline assessment.
  Participants will receive a 3-day training in their home that will include basic tablet/internet training and training on the features of the system. The training will also encompass a module on internet etiquette and security against potential spam and fraud. Participants will be provided with practice tasks in between sessions. Participants will be provided with a "hands-on" performance assessment at the end of the second session and concepts/procedures that are problematic will be reviewed.
  Interventions: Behavioral: Project 2, Phase 2: Intelligent Adaptive System
- Project 2 - Phase 2: Waitlist Control (Active Comparator): Participants will receive a 3-day training in their home. Participants will also receive a tablet, internet support for 12 months and training. This will include instructions for accessing content pertaining to the research study.
  Interventions: Behavioral: Project 2, Phase 2: Intelligent Adaptive System
- Project 3 - Phase 1: Problem Space Specification and Task Selection (No Intervention): Both the subject matter experts and older adult participants will participate in individual structured interviews for each activity category, 1.5 - 2 hours in length. This qualitative data will provide rich contextualized information regarding the specific needs of older adults for access to services, financial health management, and Medicare.gov services utilization. This data will be used to identify current barriers and facilitators to successful healthcare management that could be targeted by technology solutions and/obtain details of the challenges that are common in each activity category.
- Project 3 - Phase 2: Development of Digital Assistant Tools (No Intervention): The study includes one session that will last approximately 2 - 3 hours. The study involves interactions with digital assistants developed by the research team, the participants will answer structured interview questions regarding their experiences using the system. The researchers will assess the participants' comments along dimensions such as type of information requested, preference for format of information, points of confusion, and likes and dislikes of features, which will form the basis for a prioritized list of features/functions to be modified for the next prototype iteration.
- Project 3 - Phase 3: DATA Condition (Experimental): Participants in the DATA condition, instead of access to a generic digital assistant, will have DATA at their disposal to solve the queries and will be encouraged to use it as the primary resource. Qualitative data on how they use this tool, in isolation and in conjunction with other sources of information, will be collected. Following completion of the problems, as in Phase 2, measures of DATA usability will be collected including usefulness and comprehension associated with each tool, perceived mental workload, and usability with an efficient, two-item test based on the widely used System Usability Scale: UMUX-LITE). The investigators will then conduct an audio-recorded semi-structured exit interview about various perceptions participants had regarding the challenges associated with successfully solving the health-management problems.
  Interventions: Behavioral: Project 3, Phase 3: Intelligent Decision Support Tool
- Project 3 - Phase 3: Usual-Tool Control Condition (Active Comparator): Participants will have access to a generic, non-adapted voice assistant available on a provided tablet. The experimenter will use a standard script that allows for guidance to participants in searching for information relevant to the problems. Participants will indicate when they are ready to move on to the next problem, which will be followed by their assessment of the confidence they have in having solved the problem, their comprehension of the information associated with the problem, their assessment of the usefulness of the available information, and the perceived mental workload they experienced in solving the problem. Investigators will track, code, and analyze participants' online interactions with any websites they use. For each of the three task activity domains, overall performance scores will be computed, as will performance scores for the simpler and more complex problems.
  Interventions: Behavioral: Project 3, Phase 3: Intelligent Decision Support Tool

INTERVENTIONS:
Behavioral: Project 1, Phase 2: VR Program for Social, Activity, and Cognitive Engagement — The investigators will apply a systematic approach to the design and evaluation of an immersive Cognitive Activity Social Technology (CAST) VR intervention (using the Oculus Quest 2), that provides aging adults a suite of virtual cognitive, social, and activity engagement applications. The program will allow for virtual interactions (one-on one or groups), cultural, creativity, and educational opportunities, and gaming.
  Arms: Project 1 - Phase 2: Tablet Control Condition; Project 1 - Phase 2: VR Program
Behavioral: Project 2, Phase 2: Intelligent Adaptive System — An innovative intelligent adaptive software package aimed at providing social and cognitive support to older adults with MCI. The system will be designed to adapt to the needs and abilities of the user.
  Arms: Project 2 - Phase 2: Active Intervention Group; Project 2 - Phase 2: Waitlist Control
Behavioral: Project 3, Phase 3: Intelligent Decision Support Tool — An innovative intelligent decision tool for health decisions aims at providing health management support for older adults with and without MCI.
  Arms: Project 3 - Phase 3: DATA Condition; Project 3 - Phase 3: Usual-Tool Control Condition

SUMMARY:
Project 1: The goal of this research project is to examine usability and acceptance of virtual reality (VR) applications and their efficacy with older adults. This highly innovative cross-site Stage 1 Intervention Development Project (NIH (National Institutes of Health) Stage Model) will apply the CREATE systematic approach to the design and evaluation of an immersive VR program, Cognitive Activity Social Technology (CAST), for older adults. The program will provide a suite of virtual cognitive, social and activity engagement applications; and allow for virtual interactions.

Project 2: The goal of this Stage 1 (NIH Stage Model) Intervention Development cross-site project is to develop, using a user-centered design approach, and evaluate an innovative intelligent adaptive software package aimed at providing cognitive and social support and engagement to older adults with mild cognitive impairment (MCI). The system will be designed to adapt to the needs and abilities of the user. The investigator's goal is to develop a unique and highly innovative technology tool that can provide adaptive support to aging individuals with MCI, even as cognition might deteriorate further. Speech data collected as part of an embedded reminiscence feature will advance fundamental knowledge of how speech and language production data might serve as an early indicator of cognitive decline.

Project 3: The goal for this project is to support the cognitive components of older adults' health-management activities through development of digital assistant technology tools tailored to three exemplar healthcare management task activities: accessing support services, managing healthcare finances, and using the health-management tools provided by Medicare.gov. This project will leverage the machine-intelligence expertise of the research investigators collaborators and the research investigators experience in developing and evaluating technologies for supporting the health and wellbeing needs of older adults to harness technology to provide cognitive support to aging adults, including those with Mild Cognitive Impairment (MCI) and lower SES. The project will be comprised of three phases.

DETAILED DESCRIPTION:
Deployment of technology in healthcare and day-to- day activities is increasing and advances in technology such as artificial intelligence (AI) are increasingly aimed at supporting older adults. Yet, aging adults are often ignored in design, and robust research evaluating the usability, safety, and efficacy of these systems with older adults is limited. Even among older technology adopters, rapid changes in technology pose challenges in terms of the constant need for adaptation and continual learning. Further, there remains a lag in uptake among many older adult sub-groups, including ethnic minorities, older cohorts, those of lower socio-economic status, those living in a rural location, or with a cognitive impairment such as Mild Cognitive Impairment (MCI) or Alzheimer's Disease/Alzheimer's Disease Related Dementias (AD/ADRD). The goal of CREATE V is to harness the potential benefits and power of technology to maintain, support, and foster the cognitive, emotional, and physical health of aging adults to enhance independence, well-being, and quality of life. Given that age represents a significant risk factor for cognitive impairments such as MCI and AD/ADRD, and the criticality of cognition to everyday functioning, a thrust of the research investigators planned research is on using emerging technologies to help maintain cognitive health and provide support for those with cognitive impairments. CREATE V has a fresh vision, a focus on emerging technologies, expanded research teams, new populations such as those with cognitive impairments, and technological capabilities.

Project 1: Phase 1, akin to NIH Stage 1a, will involve usability testing across the three CREATE sites with older adults, and heuristic analysis to gather information on user preferences, usability problems, implementation, and training protocols.

Phase 2, akin to NIH Stage 1b, will involve a cross-site pilot randomized trial with a large and diverse sample of aging adults. Participants will be randomized, following a baseline assessment, to the VR CAST condition or a tablet control condition, where participants will be exposed to similar context in 2d (e.g., online museum tours). Following training on the VR program/tablet, they will use the VR program/tablet in their home for two months. The battery of measures will be re-administered at 1 and 2-months post randomization. Research investigators will collect real time data on use of the VR program/tablet. The planned project will yield significant and timely information on the feasibility of using VR support for older adults, delineate potential mediator and moderators of the benefits of VR, and design guidelines for VR interventions for older adults.

Project 2: Phase 1 of the project will yield important information on the feasibility of using technology-based approaches to support everyday activities and cognition for persons with MCI and insight on barriers to the implementation of technology-based interventions. The investigators will also gain understanding of the challenges aging adults with MCI encounter in everyday activities.

In phase 2, akin to Stage 1b, the study will involve pilot testing to evaluate the feasibility, acceptability, and usability of the system (primary outcomes) with a diverse sample of individuals with MCI at each site. Investigators will gather preliminary data on efficacy of the system with respect to secondary outcomes such as cognition, perceptions of memory functioning, social connectivity, social support, loneliness, technology proficiency, and the performance of everyday tasks. Investigators will collect real time data on system use and system adaptations. Investigators will examine potential negative consequences of use of the system, such as decreases in social networks or interactions or negative changes in life space. All assessments will occur in the participants' living environment by trained research assistants. An assessor other than the one who conducted the baseline assessment, will conduct follow-up assessments to minimize bias (i.e., assessors will be blinded to treatment condition).

Project 3: Phase 1 will use a multimethod approach across the three study sites to assess the demands and challenges facing diverse older adults in the performance of the three health- management activities. Techniques include structured focus groups of subject matter experts, cognitive task analysis of existing tools, and process tracing of older adults' task performance.

In Phase 2, investigators will use the knowledge derived from Phase 1, together with an understanding of older adults' cognitive capabilities and limitations, and their needs and preferences, to conduct iterative design of the digital assistant tools and evaluate their effectiveness and perceived usability using older adults with and without cognitive impairments and diverse in technology skills.

In Phase 3, investigators will do a comparative assessment of the digital assistant tools for the three health-management activities (4 problems in each domain) by randomizing a cross-site sample of 240 participants, with and without MCI, varying in age, ethnicity/race, SES, and technology experience, to novel tool and control conditions, assessing efficacy and usability of the novel tools. The project will yield important information on how best to design technology aids to provide cognitive support for health decision making.

Outcome measures for Projects 2 and 3 will be determined based on the conclusion of Project 1.

ELIGIBILITY:
Inclusion Criteria:

Project 1:

* 65+ years of age
* Able to read English at the 6th grade level
* Have 20/60 vision with or without correction.

Project 2:

* 62+ years of age
* Able to read English at the 6th grade level
* Have 20/60 vision with or without correction.
* Clinical diagnosis of mild cognitive impairment (MCI)
* Subjective cognitive complaints
* Evidence by clinical evaluation
* Clinical Dementia Rating Global scale of 0.5-2.0
* Probable MCI
* Montreal Cognitive Assessment (MoCA) score of 18-26
* No major Instrumental activities of daily living (IADL) impairments
* Geriatric Depression Scale of 4 or Below
* No diagnosis of dementia

Project 3:

* 60+ years of age
* Able to read English at the 6th grade level
* Have 20/60 vision with or without correction.
* MoCA score of 23 or lower

Exclusion Criteria:

All Projects:

* Blind or have visual impairments that limit their ability to view the technology.
* Deaf or have hearing impairments that limit their ability to answer telephone queries.
* Have a life-limiting/terminal illness
* Severe motor impairment (e.g., severe tremors or debilitating arthritis in their hands) that impairs ability to speak or use dominant hand

Project 1:

- Chronic neck pain/injury that might make the headset uncomfortable

Project 2:

- Cognitive impairment (MOCA ≤ 25)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1202 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Project 1, Phase 2: Perceived System Feasibility of the CAST Program as measured by the number of days used | Baseline through 2 months
  The CAST system or tablet feasibility will be assessed by evaluating participants' perception of the features of the system. Real time measures of the CAST system or tablet use will be evaluated, by the number of days used starting from baseline through two months. Measure is to be developed based on phase 1 of the study.
Project 1, Phase 2: Perceived System Feasibility of the CAST Program as measured by the number of times used per day | Baseline through 2 months
  The CAST system or tablet feasibility will be assessed by evaluating participants' perception of the features of the system. Real time measures of the CAST system or tablet use will be evaluated, using the sum of times the system was used per day or the average starting from baseline through two months. Measure is to be developed based on phase 1 of the study.
Project 1, Phase 2: Perceived System Feasibility of the CAST Program as measured by the number of features used per day | Baseline through 2 months
  The CAST system or tablet feasibility will be assessed by evaluating participants' perception of the features of the system. Real time measures of the CAST system or tablet use will be evaluated, by number of features used per day, using the sum of numbers of features used per day or the average starting from baseline through two months. Measure is to be developed based on phase 1 of the study.
Project 1, Phase 2: Mean Difference of Perceived Ease of Use of the CAST Program Assessed using the Perceived Ease of Use Questionnaire | Post-Randomization at Month 1 and Month 2
  Utilizing a 12-item scale (Perceived Ease of Use Questionnaire) which includes two subscales (perceived usefulness and perceived ease of use) with Likert response scales ranging from. 1 (Strongly disagree) - 10 (Strongly agree). The responses to the items are summed for each of the subscales. To assess ease of use, the investigators will evaluate responses to the perceived ease of use subscale. Higher sores indicate perceived ease of use of the CAST program.
Project 1, Phase 2: Mean Difference of Perceived System Usefulness of the CAST Program, assessed using the Perceived Usefulness Questionnaire | Post-Randomization at Month 1 and Month 2
  Utilizing a 12-item scale (Perceived Usefulness Questionnaire) which includes two subscales (perceived usefulness and perceived ease of use) with Likert response scales ranging from. 1 (Strongly disagree) - 10 (Strongly agree). Higher sores indicate perceived system usefulness of the CAST program. The responses to the items are summed for each of the subscales.
Project 1, Phase 2: Mean Difference in Score of CAST Program Intervention Workload, assessed using the NASA Tax Load Index (TLX) Measure | Post-Randomization at Month 1 and Month 2
  The TLX is a measure of perceived workload that assesses six dimensions of workload: Mental, Physical, and Temporal Demands, Frustration, Effort, and Performance. Administering the TLX involves two steps. First, a participant reflects on the task they're being asked to perform and looks at each paired combination of the six dimensions to decide which is more related to their personal definition of workload as related to the task. This results in a user considering 15 paired comparisons. For example, they need to decide whether Performance or Frustration "represents the more important contributor to the workload for the specific task recently performed." The second step involves participants rating each of the six dimensions on scales from Low to High or from Good to Poor. The raw score for each of the six items is multiplied by the weight from step 1 to generate the overall workload score per task.
  NASA TLX -- Scores Range from 0 (low work load) - 100 (very high work load)
Project 1, Phase 2: Mean Difference in Score of Perceived CAST Program system enjoyment Assessed using The User Experience Questionnaire | Post-Randomization at Month 1 and Month 2
  The User Experience Questionnaire. A 23-item scale that measures enjoyment and immersion of a virtual reality experience. Eleven items are related to enjoyment - these items will be summed to assess enjoyment, Scores range from 0-11, with 11 indicating greater enjoyment.
Project 2, Phase 2: Perceived System Usability of the CAST Program as Measured by the number of times used per day | Baseline through 6 months
  The CAST system or tablet usability will be assessed by evaluating participants' perception of the features of the system. Real time measures of the CAST system or tablet use will be evaluated, by the number of days used using the sum of times the system was used per day or the average, starting from baseline through six months. Measure is to be developed based on phase 1 of the study.
Project 2, Phase 2: Perceived System Usability of the CAST Program as measured by the number of times the system was used per day | Baseline through 6 months
  The CAST system or tablet usability will be assessed by evaluating participants' perception of the features of the system. Real time measures of the CAST system or tablet use will be evaluated, using the sum of times the system was used per day or the average starting from baseline through six months. Measure is to be developed based on phase 1 of the study.
Project 2, Phase 2: Perceived System Usability of the CAST Program as measured by the number of features used per day | Baseline through 6 months
  The CAST system or tablet usability will be assessed by evaluating participants' perception of the features of the system. Real time measures of the CAST system or tablet use will be evaluated, by number of features used per day, using the sum of numbers of features used per day or the average starting from baseline through six months. Measure is to be developed based on phase 1 of the study.
Project 2, Phase 2: Perceived Ease of Use of the CAST Program, assessed using the Perceived Ease of Use Questionnaire | 6 months post intervention
  Utilizing a 12-item scale (Perceived Ease of Use Questionnaire) which includes two subscales (perceived usefulness and perceived ease of use) with Likert response scales ranging from. 1 (Strongly disagree) - 10 (Strongly agree). The responses to the items are summed for each of the subscales. To assess ease of use, the investigators will evaluate responses to the perceived ease of use subscale.
Project 2, Phase 2: Perceived System Usefulness of the CAST Program, assessed using the Perceived Usefulness Questionnaire | 6-months post intervention
  Will assess participants' perception of technology-based intervention usefulness. Utilizing a 12-item scale (Perceived Usefulness Questionnaire) which includes two subscales (perceived usefulness and perceived ease of use) with Likert response scales ranging from. 0 (Strongly disagree) - 4 (Strongly agree). Higher sores indicate perceived ease of use of the CAST program. The responses to the items are summed for each of the subscales.
Project 2, Phase 2: Mean scores of participants' perception of CAST program usability and usefulness, assessed using the Usability Metric for user Experience (UMUX-Lite) questionnaire | 6-months post intervention
  Will assess participants' perception of technology-based intervention ease of use and usefulness. The Usability Metric for User Experience (UMUX-Lite) is a two-item Likert scale used for the subjective assessment of an application's perceived usability. On a 7- point scale, with 0 being strongly disagree and 6 being strongly agree, higher scores are reflective of a greater satisfaction with the system. The scoring range is from 0 to 14. A higher accumulated score is representative of a higher perception of usability.
Project 3, Phase 1: Qualitative interview assessment regarding Healthcare Challenges | During one-time condition session at Baseline Assessment
  Analysis of interview transcripts will identify common themes that will be the target of technology-based support. The general script for interviews with older adults will start with a) demographics and medical history; (b) health management strategies - current approaches for monitoring and managing chronic conditions and maintaining general wellness; (c) current use, awareness of, openness to, and concerns about technologies for health management; (d) general challenges experienced and barriers to successful health management. Investigators will then have sections of the interview script tailored to the three activity categories: access to services; financial health management, and Medicare utilization.
Project 3, Phase 3: Mixed-method assessment of usability challenges assessed using the Usability Metric for User Experience (UMUX-LITE) | During one-time condition session at Baseline Assessment
  User testing will have participants "think aloud" as they solve healthcare problems, and data will be coded for frustration and specific challenges experienced. The investigators will also use classic usability measures, for example, UMUX-LITE. The Usability Metric for User Experience (UMUX-Lite) is a two-item Likert scale used for the subjective assessment of an application's perceived usability. On a 7 point scale, with 0 being strongly disagree and 6 being strongly agree, higher scores are reflective of a greater satisfaction with the system.
Project 3, Phase 3: Comprehension and Decision Making Accuracy | During one-time condition session at Baseline Assessment
  For hypothetical healthcare challenges participants will be presented with, they will afterward be tested on their comprehension of important terms, and their decision-making accuracy will be evaluated, for participants with and without access to novel technology tools developed as part of this project. The comprehension and decision making accuracy measure is to be developed based on projects 1 and 2 of the study.

SECONDARY OUTCOMES:
Project 1, Phase 2: Mean Difference in Score of Social Support and Connectivity Assessed using The Social Connectedness Measure | Post-Randomization at Month 1 and Month 2
  Scales used to measure two aspects of social isolation: social disconnectedness and perceived isolation, as well as perceived availability of social support.
  The Social Connectedness measure is a 15 item scale consisting of 3 sections with different likert response scale. Section 1 is a 4 item scale ranging from 0 - 5 points (20 total points). Section 2 is a 6-item scale ranging from 1 - 3 points (18 total points). Section 3 is a 5-item scale ranging from 1 - 5 points (25 total points). For Section 1, a higher score is reflective of increased connectedness while for Section 2 and 3, a higher score is a reflective of a higher level of disconnectedness. For sections 1-3, a mean difference in score will be calculated.
Project 1, Phase 2: Mean Difference in Score of Quality of Life, assessed using The Quality of Life Questionnaire | Post-Randomization at the Baseline assessment, Month 1 and Month 2
  Will assess the participant's quality of life by having the participant rate different aspects of their life using one of four words: poor, fair, good, or excellent. They are instructed to think about different aspects of their life, like physical health, energy, family, money, and others to assess their situation in each area.
  The Quality of Life questionnaire is a 13-item scale with Likert response scales ranging between 1 and 4 points. The measure's total score can range between 13 - 52 points. A higher total score is reflective of a higher quality of life while a lower score is reflective of a poorer quality of life.
Project 1, Phase 2: Mean Difference in Score of reported depression, assessed using the Center for Epidemiological Studies-Depression (CES-D) Scale | Post randomization at the baseline assessment, month 1 and month 2.
  The CES-D is a self-report depression scale for research in general population. It is a 20 item questionnaire consisting of likert response scales ranging from 0-3 points. The total score range is 0 - 60 points. Higher scores indicate participants have a greater level of self reported depression.
Project 1, Phase 2: Mean Difference in score of participants self-reported health, assessed using the 36-Item Short Form Health Survey questionnaire (SF-36 Short Form) | Post randomization at the baseline assessment, month 1 and month 2.
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability. The 8 subscales or domains are as follows:
  Physical functioning (10 items);
  Role limitations due to physical health (4 items); Role limitations due to emotional problems (4 items); Energy/fatigue (4 items); Emotional well-being (5 items); Social functioning (2 items); Pain (2 items); General health (5 items).
Project 2, Phase 2: Mean Difference in Score of Social Support and Connectivity Assessed using The Social Connectedness Measure | Baseline and 6 month post intervention
  Scales used to measure two aspects of social isolation: social disconnectedness and perceived isolation, as well as perceived availability of social support.
  The Social Connectedness measure is a 15-item scale consisting of 3 sections with different likert response scale. Section 1 is a 4-item scale ranging from 0 - 5 points (20 total points). Section 2 is a 6-item scale ranging from 1 - 3 points (18 total points). Section 3 is a 5-item scale ranging from 1 - 5 points (25 total points). For Section 1, a higher score is reflective of increased connectedness while for Section 2 and 3, a higher score is a reflective of a higher level of disconnectedness. For sections 1-3, a mean difference in score will be calculated.
Project 2, Phase 2: Mean Difference in Score of Quality of Life, assessed using The Quality of Life Questionnaire | Baseline and 6 month post intervention
  Will assess the participant's quality of life by having the participant rate different aspects of their life using one of four words: poor, fair, good, or excellent. They are instructed to think about different aspects of their life, like physical health, energy, family, money, and others to assess their situation in each area.
  The Quality of Life questionnaire is a 13-item scale with Likert response scales ranging between 1 and 4 points. The measure's total score can range between 13 - 52 points. A higher total score is reflective of a higher quality of life while a lower score is reflective of a poorer quality of life.
Project 2, Phase 2: Mean Difference in Score of reported depression, assessed using the Center for Epidemiological Studies-Depression (CES-D) Scale | Baseline and 6 month post intervention
  The CES-D is a self-report depression scale for research in general population. It is a 20 item questionnaire consisting of likert response scales ranging from 0-3 points. The total score range is 0 - 60 points. Higher scores indicate participants have a greater level of self reported depression.
Project 2, Phase 2: Mean Difference in score of participants self-reported health, assessed using the 36-Item Short Form Health Survey questionnaire (SF-36 Short Form) | Baseline and 6 month post intervention
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability. The 8 subscales or domains are as follows:
  Physical functioning (10 items); Role limitations due to physical health (4 items); Role limitations due to emotional problems (4 items); Energy/fatigue (4 items); Emotional well-being (5 items); Social functioning (2 items); Pain (2 items); General health (5 items).
Project 2, Phase 2: Mean Difference in scores of participants' perceived memory function, assessed using the Perception of Memory Function questionnaire | Baseline and 6 month post intervention
  The Perception of Memory Function Questionnaire is a self-report questionnaire for clinicians and researchers to use for assessing metamemory in middle-aged and older adults. It consists of 64 items to be rated on a 7-point Likert scale; the items load on four factors, each of which associated with a specific aspect of memory. The 7-point scale ranges from major problems (1) to no problems (7). Participants on the lower end of the scoring range indicate experiencing more memory problems.
Project 3, Phase 3: Comprehension and Decision Making Tool Usability | During one-time condition session at Baseline Assessment
  The Comprehension and Decision making tool will measure participants' perception of technology-based intervention ease of use and usefulness. The Comprehension and Decision making tool measure is to be developed based on projects 1 and 2 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Czaja, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Florida State University, Tallahassee, Florida
  - University of Illinois Urbana-Champaign, Champaign, Illinois
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan for resource sharing is based on the National Institutes of Health/National Institute on Aging (NIH/NIA) Data Sharing Policy. The investigators plan, consistent with the NIH goals of data sharing, is to promote use of the rich CREATE database by the larger research community as this will further the impact of CREATE and expand possibilities for collaboration. It will also allow other researchers to expedite the translation of the research findings into knowledge, products, and procedures. Further, the plan is devised to make the data as widely and freely available as possible while at the same time safeguarding the privacy of participants and protecting confidential and proprietary data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data from research projects will be made available no later than acceptance of publication of the main findings from the final data set. There is no end date to access the data from the research projects.
Access Criteria: The investigators agree to share the data with researchers working under an institution with Federal Wide Assurance who agree to a data sharing agreement that stipulates protection of participant privacy and data confidentiality, acknowledgement of CREATE, that the data will be used for research purposes only, and that the data will not be transferred to other users. The computerized data will include raw data, derived variables, all necessary documentation as described in the National Archive of Computerized Data on Aging depositor agreement. All data will be de-identified. The investigators will follow the guides published by the US Department of Health and Human Services in this respect. Each data set will include data documentation to ensure that others can use the data set and to minimize confusion. Information about where and how to locate and access the data will be available in any publications and presentations authored by CREATE investigators.
URL: https://create-center.ahs.illinois.edu/